CLINICAL TRIAL: NCT02492776
Title: A Study in Healthy Subjects to Assess the Multiple-Dose Pharmacokinetics of Two AF-219 Formulations
Brief Title: A Multiple-Dose Pharmacokinetics Study of Two Gefapixant (AF-219/MK-7264) Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7264-020; AF219-020 (Other: Afferent Pharmaceuticals)
Record Dates: First submitted 2015-06-15; First posted 2015-07-09 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Omeprazole; Gefapixant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefapixant + Omeprazole (Experimental): Gefapixant oral tablets (25mg, 50 mg) administered twice daily for 13 days + Omeprazole oral capsules (20 mg) administered once daily for 8 days
  Interventions: Drug: Omeprazole; Drug: Gefapixant

INTERVENTIONS:
Drug: Omeprazole — 20 mg oral capsules administered once daily for 8 days
  Other Names: Prilosec
Drug: Gefapixant — Gefapixant oral tablet (25 mg administered as a divided 50 mg tablet) administered twice daily for 5 days
  Other Names: AF-219; MK-7264
Drug: Gefapixant — Gefapixant oral tablet (50 mg tablet) administered twice daily for 8 days
  Other Names: AF-219; MK-7264

SUMMARY:
The purpose of this study is to compare the multiple dose pharmacokinetics (PK) of two gefapixant (AF-219) formulations; to assess the effect of omeprazole on the multiple dose PK of two gefapixant formulations; and, to assess the safety and tolerability of gefapixant.

ELIGIBILITY:
Inclusion Criteria:

* Must be informed of the nature of the study and have provided written informed voluntary consent;
* Able to speak, read, and understand English;
* Healthy males or females, of any race, between 18 and 55 years of age, inclusive;
* Body mass index (BMI) >18.5 and <32.0 kg/m2 and weigh 50 - 100 kg;
* In good general health;
* Non-smokers or intermittent (social) smokers for at least 5 years, and able to refrain from smoking (or using nicotine) while in confinement;
* If a female of child-bearing potential (i.e., have not undergone a hysterectomy or bilateral oophorectomy) or not post-menopausal (defined as no menses for at least 12 months), agree to use 2 forms of acceptable birth control; or if a male, they and/or their partner of child-bearing potential agree to use 2 forms of acceptable birth control; when in line with the preferred life style of the subject, true and complete abstinence (not periodic abstinence) is acceptable;

Exclusion Criteria:

* Any disease or condition that might affect drug absorption, metabolism, or excretion or clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease;
* Clinically significant illness or clinically significant surgery within 4 weeks before the administration of study medication;
* Any past sinus surgery, upper respiratory tract infection within 2 weeks before dosing, or history of hay fever during the time of the year that dosing will be taking place;
* History of GERD, heartburn, or nausea more than once a month, or any similar symptoms requiring the regular use of antacids, or any use of H2 histamine blockers or proton pump inhibitors within 12 months of Screening;
* Have a positive screening test for Helicobacter pylori;
* QTcB >450 msec in males or >470 msec in females;
* Known or suspected hypersensitivity or allergic reaction to any of the components of gefapixant or omeprazole capsules;
* If female, is pregnant or breast feeding, or has a positive pregnancy test pre dose;
* Blood loss or blood donation of >550 mL within 90 days or plasma donation >500 mL within 14 days before administration of the first dose of study drug;
* Chronic use of any systemic medications (other than allowable oral and implanted contraceptives and with the exception of vitamins taken at standard supplement doses); use of a drug therapy (including herbal preparations, e.g., St. John's wort) known to induce or inhibit hepatic drug metabolism within 30 days before the first dose of study medication; or use of any medications [prescription or over the counter (OTC)], including antacids, high dose multivitamins, nutritional supplements, and herbal preparations, within 14 days before the first dose of study drug;
* Past or current history or evidence of drug or alcohol abuse, regular use of more than 2 units of alcohol per day (1 unit of alcohol = 150 mL of wine, 360 mL of beer, or 45 mL of alcohol 40%), use of any recreational soft drugs (e.g., marijuana) within 3 months of screening, use of any hard drugs (such as cocaine, phencyclidine (PCP), and crack) within 1 year of screening, and/or a positive screen for substances of abuse or alcohol at screening or pre dose;
* Ingestion of grapefruit or grapefruit juice within 48 hours before dose administration;
* Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C antibody, or human immunodeficiency virus (HIV) antibody;
* Receipt of an investigational product or device, or participation in a drug research study within a period of 30 days (or 5 half lives of the drug, whichever is longer) before the first dose of study medication;
* Receipt of an investigational immunomodulator or monoclonal antibody within 180 days (or 5 half lives, whichever is longer) before the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2015-08-04 (Actual); Study Completion 2015-08-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentration profiles of two different oral formulations of gefapixant | 12 hours
  Plasma gefapixant concentration versus time profiles will be plotted for each subject; similar summary plots will be constructed for each treatment period. Plasma gefapixant PK parameters will be calculated using noncompartmental methods and summarized using descriptive statistics by each treatment.
Plasma concentration profile of gefapixant following administration of omeprazole | 5.5 hours
  Analysis of variance (ANOVA) will be performed on log normal-transformed Cmax and AUC0-t values to determine the extent of a drug interaction, if any, of omeprazole on the plasma gefapixant PK parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Swearingen, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

REFERENCES:
- [Result] Gupta P, Hussain A, Ford AP, Smith S, Nussbaum JC, Stoch A, Iwamoto M. Clinical Formulation Bridging of Gefapixant, a P2X3-Receptor Antagonist, for the Treatment of Chronic Cough. Clin Pharmacol Drug Dev. 2022 Sep;11(9):1054-1067. doi: 10.1002/cpdd.1105. Epub 2022 May 5. PMID 35510785